CLINICAL TRIAL: NCT01147211
Title: A Phase I Dose Defining Study For MK-2206 Combined With Gefitinib In NSCLC Population Enriched With EGFR Mutation
Brief Title: Dose Defining Study For MK-2206 Combined With Gefitinib In Non Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201001017M
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: dose defining; MK-2206; NSCLC With EGFR Mutation; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK2206 in combination with Gefitinib (Experimental): MK-2206 will be administered orally in a starting dose level of 135 mg on a schedule of Qwk in repeating 3-week treatment cycles in combination with gefitinib in continuous 21-day cycles for the duration of the study
  Interventions: Drug: MK2206

INTERVENTIONS:
Drug: MK2206 — MK-2206 will be administered orally in a starting dose level of 135 mg on a schedule of Qwk in repeating 3-week treatment cycles in combination with gefitinib in continuous 21-day cycles for the duration of the study

SUMMARY:
This is a phase I study of MK2206 (an AKT inhibitor)and gefitinib in nonsmall cell lung cancer patients who failed prior chemotherapy and epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI). The patient population is enriched for EGFR mutations.

The purpose of this study is to determine whether it is safe to administered MK-2206 in combination with gefitinib in adult patients with locally advanced or metastatic non-small cell lung cancer. The second purpose of this study is to define the MTD (Maximum Tolerated Dose) of MK-2206 when combined with gefitinib.

A standard 3-3 dose escalation scheme of MK-2206 with fix dose gefitinib is used in this study.

DETAILED DESCRIPTION:
Preclinical data from communication with Merck clinical and pre-clinical group support the application of MK2206 and an EGFR-TKI, and the synergistic effect of this combination. This proposed study is a phase I dose defining study to define the MTD (Maximum Tolerated Dose) of MK-2206 when combined with gefitinib.

MK-2206 is a potent, orally active, allosteric inhibitor of human AKT1, AKT2, and AKT3 with preclinical anti-tumor activity.

This is a Phase I, single-center, open-label, non-randomized, dose-escalation study in patients with locally advanced or metastatic NSCLC. Patients who previously failed and progressed through EGFR inhibitor such as erlotinib or gefitinib and up to one line of chemotherapy will be enrolled into the study. Patients will be administered with oral MK-2206 and a standard dose of EGFR inhibitor gefitinib.

This study will be conducted in three cohorts to identify a recommended Phase II dose (RP2D) of MK-2206 in combination with standard dose of gefitinib (250 mg QD). Cohorts of 3 patients will be enrolled sequentially on escalating doses of MK-2206 administered in combination with a standard dose of gefitinib. Patients will advance doses of MK2206 if 0/3 patients or 0-1/6 develop DLT (Dose-Limiting Toxicity). If 1/3 patient develops DLT, the cohort will be expanded to 6. If 2/6 patients developed DLT, the dose will be de-escalate to 90 mg Qwk. The highest dose cohort with 0-1/6 with DLT will be deemed as MTD and used as cohort expansion for a total of 15 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically-confirmed locally advanced or metastatic NSCLC who have received EGFR inhibitors (such as gefitinib, erlotinib) for at least 3 months and progressed and also received at least one line of platinum-based chemotherapy. In the MTD expansion cohort, patients must have documented progression on gefitinib, erlotinib, afatinib(BIBW2992) or PF299804 within 4 weeks of starting gefitinib and MK2206 treatment. There should be no anticancer treatment between above mentioned treatment and protocol treatment.
2. Patient is male or female and ≥ 20 years of age on the day of signing informed consent.
3. Patient must have performance status ≤ 2 on the ECOG Performance Scale.
4. Patient must have adequate organ function
5. Female patient of childbearing potential has a negative serum or urine pregnancy test β-hCG within 72 hours prior to receiving the first dose of study medication.
6. Patient have completed any targeted therapy (excluding gefitinib, erlotinib or any small molecule EGFR tyrosine kinase inhibitors ), any chemotherapy regimens and therapeutic radiation for a minimum of 30 days prior to starting of treatment, and palliative radiotherapy covering less than 30% bone marrow for a minimum 14 days prior to starting of treatment.
7. Prior usage of BIBW2992 are allowed if patient failed on BIBW2992 over 3-month therapy.
8. Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent.
9. Patient is able to swallow capsules and has no surgical or anatomical condition that will preclude the patient from swallowing and absorbing oral medications on an ongoing basis.

Exclusion Criteria:

1. Patient who has had chemotherapy, radiotherapy, biological therapy, or BIBW2992 (except gefitinib, erlotinib) within 30 days (6 weeks for nitrosoureas, mitomycin C or bevacizumab), or 5x half-life, whichever is longer, prior to starting of treatment, or who has not recovered from the adverse events due to previous agents administered more than 30 days prior to Study Day 1. If the patient has residual toxicity from prior treatment, toxicity must be ≤ Grade 1.
2. Patients who has had major surgery within 4 weeks prior to starting of treatment or expect major surgery in the study duration.
3. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days, or 5x half-life from prior agents, whichever is longer, of Day 1 of this study.
4. Patient has known active CNS metastases and/or carcinomatous meningitis. However, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for 1 month prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis (2) off steroids or on a stable dose of steroids.
5. Patient with a primary central nervous system tumor.
6. Patient has known hypersensitivity to the components of study drug or its analogs.
7. Patient has a history or current evidence of heart disease.
8. Patient with evidence of clinically significant bradycardia (HR < 50), or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, 2nd degree AV block (Mobitz Type 2), or patients taking non-dihydropyridine calcium channel blockers, or digoxin.
9. Patient with uncontrolled hypertension (i.e. ≥160/90 mHg). Patients who are controlled on antihypertensive medication will be allowed to enter the study.
10. Patient at significant risk for hypokalemia (eg. patients on high dose diuretics, or with recurrent diarrhea)
11. Patient is a known diabetic patient
12. Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
13. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
15. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
16. Patient is known to be Human Immunodeficiency Virus (HIV)-positive
17. Patient currently has active Hepatitis.
18. Patient has symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible.
19. Patient is receiving treatment with oral corticosteroids (note: inhaled corticosteroids or premedication for chemotherapy are permitted).
20. Patient is using a potent CYP3A4 inhibitor or inducer (See Appendix 6.2) for a list of potent CYP3A4 inhibitors or inducers). Patients who have discontinued any of these medications must have a wash-out period of at least 5 days or at least 5 half-lives of the drug (whichever is longer) prior to the first dose MK-2206.
21. Patient who has received gefitinib and discontinued due to gefitinib-related toxicity.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
to provide safety assessment and define dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of MK-2206 in combination with gefitinib in NSCLC | 21 days

SECONDARY OUTCOMES:
To explore the anti-tumor activity and to assess the pharmacokinetic profile of MK-2206 in combination with gefitinib. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsin Yang, MD, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan